CLINICAL TRIAL: NCT06624215
Title: A Retrospective Multicenter Evaluation of Short-Term Outcomes After Acute Care Appendectomy
Brief Title: Retrospective Acute Care Appendectomy Study
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI MP-APP-01
Record Dates: First submitted 2024-09-03; First posted 2024-10-02 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Acute Appendicitis
Keywords: Appendectomy; Robotic-assisted; Acute care; Laparoscopic
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Robotic-assisted appendectomy subjects: Approximately 500 subjects will be enrolled in this group who have undergone an emergent or urgent robotic-assisted appendectomy for acute appendicitis in a reverse chronological order from 30 days prior to IRB approval going back to 2018.
  Interventions: Procedure: Appendectomy
- Laparoscopic appendectomy subjects: Approximately 500 subjects will be enrolled in this group who have undergone an emergent or urgent laparoscopic appendectomy for acute appendicitis in a reverse chronological order from 30 days prior to IRB approval going back to 2018.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Robotic-assisted or laparoscopic appendectomy for acute appendicitis.

SUMMARY:
The purpose of this retrospective study is to compare perioperative data for subjects who have undergone an emergent or urgent robotic-assisted or laparoscopic appendectomy for acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 22 years of age or older at time of procedure
* Subject has undergone robotic-assisted or laparoscopic emergent or urgent appendectomy for acute appendicitis between 2018 and 30 days prior to IRB approval

Exclusion Criteria:

* Subject with appendiceal neoplasms
* Subject who underwent a single-port appendectomy
* Subject who was pregnant or breastfeeding at the time of the procedure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 500 patients who have undergone laparoscopic emergent or urgent appendectomies and approximately 500 patients who have undergone robotic-assisted emergent or urgent appendectomies for acute appendicitis in a reverse chronological order from 30 days prior to IRB approval going back to 2018, will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Operative time | Intraoperative
Procedure time | Intraoperative
Conversion | Intraoperative
Adverse events | Intraoperative and postoperative out to 30 days from procedure date
Mortality rate through 30 days | Intraoperative and postoperative out to 30 days from procedure date
  All cause
Unplanned procedure-related readmission rate through 30 days | Discharge through 30 days
Concomitant procedures | Intraoperative
Estimated blood loss | Intraoperative
Severity of appendicitis | Preoperative
Unplanned procedure-related reoperation rate through 30 days | Postoperative through 30 days
Length of stay | Start of procedure to discharge from the hospital (check-out time), up to approximately one week
  Total number of days the subject stayed in the hospital after the index procedure prior to being discharged.
Discharge disposition | Discharge from the hospital (check-out time), up to approximately one week.
  Where the subject was discharged to when released from the hospital
Blood Transfusion | Intraoperative and discharge from the hospital (check-out time), up to approximately one week.
  Any occurrence of blood transfusion either at the time of the procedure or at any point during the post-procedure hospitalization until the participant is discharged.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Ohio State University, Columbus, Ohio
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - Christus Santa Rosa Health Care Corporation, New Braunfels, Texas